CLINICAL TRIAL: NCT00940849
Title: Gastric Emptying of Plant Sterol-containing Mini Drinks in Different Meal Intake Scenarios and Their Effect on Gallbladder Emptying
Brief Title: Gastric Emptying and Gallbladder Motility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: MEC 09-2-042
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Gastric Emptying

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietary Supplement: Plant sterol containing drink (Experimental): The test products used in the study will be a commercially available PS drink and a ready to eat macaroni meal
  Interventions: Dietary Supplement: Plant sterol containing drink; Dietary Supplement: Standard macaroni meal

INTERVENTIONS:
Dietary Supplement: Plant sterol containing drink — The test products used in the study will be a commercially available PS drink and a ready to eat macaroni meal
Dietary Supplement: Standard macaroni meal — The test products used in the study will be a commercially available PS drink and a ready to eat macaroni meal

SUMMARY:
Background of the study:

Plant sterols can play an important role in lowering plasma cholesterol. The extent to which plant sterols can reduce plasma cholesterol levels depends on the intake scenario. We suggest that the difference in these effects depends on gastric emptying and bile secretion.

Objective of the study:

The aim of this study is to gain insight in the mechanisms that may be involved in the effects of plant sterol drinks on gastric emptying and gallbladder motility. In order to test this, we compare the different effects of the consumption of a plant sterol containing drink prior to, during and after a standardized meal.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Sex: male
* Age: 18-55 years
* Body Mass Index (BMI): 20-25 kg/m2

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/ hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery which might limit participation in or completion of the study protocol.
* Use of any medication on regular basis.
* Use of paracetamol prior to treatment (≤ 48 hour).
* Use of plant sterol/stanol enriched products or supplements 3 months prior to the study.
* Blood donations less than three months previous to study enrolment.
* Known hypersensitivity or allergy towards paracetamol.
* Hyperlipidaemia (TG > 3 mmol/L and/or tot. chol. > 8 mmol/L)
* Corn products prior to treatment (≤ 48 hour)
* Presence of gallbladder stones.
* Known allergy for cow milk and/or lactose intolerance

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
GB volume measurement by ultrasonography | September 2009

SECONDARY OUTCOMES:
GE rate measurement by 13C stable isotope breath test and plasma paracetamol concentration by clinical chemistry analysis | December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD PhD, Principal Investigator — Maastrich University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Result] Keszthelyi D, Knol D, Troost FJ, van Avesaat M, Foltz M, Masclee AA. Time of ingestion relative to meal intake determines gastrointestinal responses to a plant sterol-containing yoghurt drink. Eur J Nutr. 2013 Jun;52(4):1417-20. doi: 10.1007/s00394-012-0440-3. Epub 2012 Aug 23. PMID 22915051